CLINICAL TRIAL: NCT03943238
Title: Phase 1 Study of Total Lymphoid Irradiation, Total Body Irradiation, Anti-Thymocyte Globulin and Purified Donor CD34+, T-cell and Recipient T Regulatory Cell Transfusion in Human Leukocyte Antigen Mismatched Living Donor Kidney Transplantation
Brief Title: TLI, TBI, ATG & Hematopoietic Stem Cell Transplantation and Recipient T Regs Therapy in Living Donor Kidney Transplantation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stanford University (Other)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other); Northwestern University (Other)
Responsible Party: Principal Investigator, Everett Meyer, Principal Investigator, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 50540
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Living Donor Kidney Transplantation
Keywords: kidney transplant; Immunological Tolerance; Tregs; Stem cells

STUDY DESIGN:
Intervention Model Description: In this phase 1 study, a conditioning regimen of Total Lymphoid Irradiation, Anti-Thymocyte Globulin and Purified Donr CD34+, T cell and Recipient T regulatory Cell Transfusion in Human Leukocyte Antigen Mismatched Living Donor Kidney Transplantation will be studied
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combined kidney/stem cell transplants and recipient's Tregs (Experimental): Preparatory regimen including TLI, TBI, ATG after kidney transplantation followed by infusion of donor CD34+, T cell and recipient Tregs
  Interventions: Biological: Infusion of Donor Hematopoetic Stem Cells and Recipient Tregs

INTERVENTIONS:
Biological: Infusion of Donor Hematopoetic Stem Cells and Recipient Tregs — Living donor kidney transplant recipients will receive after a preparatory regimen of total lymphoid irradiation, total body irradiation and anti-thymocyte globulin an infusion of purified donor CD34+ of >10 x10^6 cells /Kg, 100 x 10^6 donor T cell/ Kg and and an escalated dose of recipient Tregs starting at 25 x10^6/Kg.

SUMMARY:
This study will determine whether a preparatory regimen including total lymphoid irradiation (TLI), total body irradiation (TBI), anti-thymocyte globulin (ATG) and infusion of the donor hematopoietic stem cells when given along with recipient regulatory T cells (Tregs) will allow for eventual discontinuation of anti-rejection drugs after living donor kidney transplantation.

DETAILED DESCRIPTION:
It has been demonstrated that hematopoietic mixed chimerism or the coexistence of both donor and recipient immune cells can lead to tolerance to the graft in absence of graft versus host disease (GVHD). The goal of this pilot study is to determine if recipients of living donor kidney transplant can be successfully withdraw from immunosuppressive drugs. The patients will receive a preparatory regimen consisting of TLI and a low single dose of TBI and ATG following their kidney transplantation. Two weeks later, they will receive purified hematopoietic stem cells (CD34+) and Tcells that have been collected 6 weeks prior from their kidney donor. Regulatory T cells (Tregs) that have been collected from the recipient prior to the transplantation and expanded in vitro will be infuse the following day to enhance the chance of engraftment of the donor bone marrow cells. If chimerism develops and persists, the immunosuppressive drug will be tapered and stop. Mycophenolate mofetil (MMF) will be stopped 12 months after transplantation and if the chimerism remains stable, tacrolimus will be stopped 6 months later. The dose of Tregs will be escalated if the % of donor chimerism is not at least 25% during the first 60 days.

ELIGIBILITY:
Inclusion Criteria:

1. All consenting adults who are 18 to 65 years, living donor renal transplant recipients at Stanford University Medical Center or Northwestern Medicine who have a haplotype matched (minimum single Human Leukocyte Antigen - DR locus (HLA-DR) and HLA-A or B match) living related or unrelated donor.
2. Patients who agree to participate in the study and sign an Informed Consent.
3. Patients who have no known contraindication to administration of rabbit ATG or radiation.
4. Males and females of reproductive potential who agree to practice a reliable form of contraception for at least 1 year posttransplant

Exclusion Criteria:

1. Previous treatment with rabbit ATG or a known allergy to rabbit proteins.
2. History of malignancy with the exception of non-melanoma skin malignancies.
3. Pregnant women or nursing mothers.
4. Serological evidence of HIV, Hepatitis B surface antigen positive (HBsAg+), or Hepatitis C infection. Epstein Barr Virus (EBV) positive to EBV negative.
5. Leukopenia (with a white blood cell count < 3000/mm3) or thrombocytopenia (with a platelet count < 100,000/mm3).
6. Panel Reactive Antibody (PRA) greater than 80% or demonstration of historic and/or current donor specific antibody (DSA)
7. Prior organ transplantation
8. High risk of primary kidney disease recurrence
9. Advanced coronary or vascular disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Count of participants with sustained mixed chimerism of >25% at 18 months | Month 18
  Chimerism is defined as the co-existence of the immune cell from both the donor and the recipient.
Count of participants able to withdraw from immunosuppressive drugs without evidence of rejection at 18 months | Month 18

SECONDARY OUTCOMES:
Count of participants with adverse events associated with the infusion of the Tregs cell product | up to 2 years
Count of participants with bacterial, viral, or fungal infections | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Everett Meyer, MD, Study Director — Stanford University
Locations (2):
- United States (2):
  - Stanford University, Palo Alto, California
  - Nothwestern University, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leventhal JR, Ildstad ST. Tolerance induction in HLA disparate living donor kidney transplantation by facilitating cell-enriched donor stem cell Infusion: The importance of durable chimerism. Hum Immunol. 2018 May;79(5):272-276. doi: 10.1016/j.humimm.2018.01.007. Epub 2018 Mar 2. PMID 29409743
- [Background] Ildstad ST, Leventhal J, Wen Y, Yolcu E. Facilitating cells: Translation of hematopoietic chimerism to achieve clinical tolerance. Chimerism. 2015 Apr 3;6(1-2):33-9. doi: 10.1080/19381956.2015.1130780. Epub 2016 Jan 8. PMID 26745761
- [Background] Scandling JD, Busque S, Shizuru JA, Lowsky R, Hoppe R, Dejbakhsh-Jones S, Jensen K, Shori A, Strober JA, Lavori P, Turnbull BB, Engleman EG, Strober S. Chimerism, graft survival, and withdrawal of immunosuppressive drugs in HLA matched and mismatched patients after living donor kidney and hematopoietic cell transplantation. Am J Transplant. 2015 Mar;15(3):695-704. doi: 10.1111/ajt.13091. PMID 25693475
- [Background] Scandling JD, Busque S, Shizuru JA, Engleman EG, Strober S. Induced immune tolerance for kidney transplantation. N Engl J Med. 2011 Oct 6;365(14):1359-60. doi: 10.1056/NEJMc1107841. No abstract available. PMID 21991976
- [Background] Scandling JD, Busque S, Lowsky R, Shizuru J, Shori A, Engleman E, Jensen K, Strober S. Macrochimerism and clinical transplant tolerance. Hum Immunol. 2018 May;79(5):266-271. doi: 10.1016/j.humimm.2018.01.002. Epub 2018 Jan 9. PMID 29330112